CLINICAL TRIAL: NCT05370703
Title: A Prospective, Randomized, Open-label, Clinical Study to Evaluate the Effect of Mobile Applications "My A:Care" and "Smart Coach" on the Lipid-lowering Treatment Adherence of Subjects With Dyslipidemia in Thailand
Brief Title: A Clinical Study to Evaluate the Effect of Mobile Applications "My A:Care" and "Smart Coach" on the Lipid-lowering Treatment Adherence of Subjects With Dyslipidemia in Thailand
Acronym: My A:Care
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: EPID-I21-0159
Record Dates: First submitted 2022-04-01; First posted 2022-05-11 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Standard of Care (SOC) group: This group will continue their current lipid-lowering therapy and will not need to download any mobile application.
- SOC + My A:Care group:: This group will continue their current lipid-lowering therapy along with access to the mobile application My A:Care that supports medication adherence through motivational messages and challenges, health insights, and medication reminders.
  Interventions: Behavioral: My A:care
- SOC + Smart Coach group:: This group will continue their current lipid-lowering therapy along with access to the mobile application Smart Coach that supports medication adherence through personalized motivational messages and challenges, health insights, and medication reminders. Personalization of the messages and challenges will be based on a behavioral profiling Social, Psychological, Usage, Rational (SPUR™) questionnaire that is completed at randomization to the Smart Coach application.
  Study site will guide the subjects on how to use these mobile applications. Eligibility assessment will be based on information collected at screening/baseline visit (Visit 1) and assessment of Part 1 of MARS 5VA questionnaire. Adherence at baseline (Visit 1) and after 12 weeks of observation (Visit 2), will be evaluated by the complete MARS 5VA (Part 1 and 2) questionnaire. Each subject will be followed up for approximately 12 weeks from randomization at Visit 1.
  Interventions: Behavioral: Smart Coach

INTERVENTIONS:
Behavioral: My A:care — Mobile application with Motivational messages
  Groups: SOC + My A:Care group:
Behavioral: Smart Coach — Mobile application with Motivational messages
  Groups: SOC + Smart Coach group:

SUMMARY:
A prospective, randomized, open-label, clinical study to evaluate the effect of mobile applications "My A:Care" and "Smart Coach" on the lipid-lowering treatment adherence of subjects with dyslipidemia in Thailand

DETAILED DESCRIPTION:
This is a prospective, randomized, open-label, clinical study in subjects with dyslipidemia and suboptimal adherence to their current lipid-lowering therapy in Thailand. Suboptimal adherence is defined as having <22 points score on the Part 1 of MARS-5VA questionnaire. This questionnaire comprises 2 parts, Medication Adherence Report Scale (MARS-5) as Part 1 and two Visual Analogue Scales (VAS) as Part 2. The complete MARS-5VA questionnaire (Part 1 and 2) will be used to evaluate subject adherence to lipid-lowering therapy in the study. The Part 1 of MARS-5VA will also be used to confirm subject's eligibility at screening. Subjects who are continuing the stable lipid-lowering therapy for at least 1 month are being considered for this study. Subjects will be randomized to different types of behavior interventions using mobile applications that will be used in addition to their current standard of care (SOC) lipid-lowering therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged 18-75 years (inclusive)
2. Subjects who have provided written informed consent
3. Subjects who were diagnosed with dyslipidemia and initiated lipid-lowering therapy based on local treatment guidelines, between 9 months and 1 month prior to the screening visit
4. Subjects who were on a stable lipid-lowering therapy within 1 month prior to the screening visit
5. Subjects who are not compliant with the prescribed lipid-lowering therapy, assessed as having <22 points score on the Part 1 of MARS-5VA questionnaire at the screening visit
6. Subjects for whom lipid profile laboratory data is available from routine care within 14 days prior to the screening visit
7. Subject must have their own Android operating system smart phone and a data package suitable for the installation and running of the mobile application and sending and receiving data
8. Willing and able to operate the mobile devices, including use of all study-related smartphone applications; able to proof regular use of mobile applications in their daily life.
9. Able to read and understand Thai
10. Willing and able to comply with the study requirements.

Exclusion Criteria:

1. Subjects who are diagnosed with myocardial infarction or stroke or unstable angina within 2 months prior to screening, subjects who are hospitalized for their cardio-vascular condition and requiring changes in administration of their lipid-lowering medication
2. Subjects who experienced undesirable effects of their lipid-lowering medication and who might, in the opinion of the investigator, require its modification or discontinuation during the 12 weeks of observation period of the study
3. Subjects receiving injectable lipid-lowering therapy
4. Subjects who are currently using other medication-use-related mobile applications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective, randomized, open-label, clinical study in subjects with dyslipidemia and suboptimal adherence to their current lipid-lowering therapy in Thailand.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-04-26 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2022-11-18 (Actual)

PRIMARY OUTCOMES:
Impact of mobile applications (My A:Care and Smart Coach) on adherence to the lipid-lowering therapy in subjects with dyslipidemia using MARS-5VA questionnaire | 12 weeks (± 7 days)
  Adherence is measured by change from Baseline in MARS-5VA Scores at 12 Weeks

SECONDARY OUTCOMES:
Impact of mobile applications (My A:Care and Smart Coach) on level of lipid control in subjects with dyslipidemia by measuring the subject's lipid profile | 12 weeks (± 7 days)
  Level of lipid control is measured by change from Baseline in the subject's lipid profile at 12 weeks
Impact of mobile applications (My A:Care and Smart Coach) on the subjects' perception to medications in general using BMQ-General-12 and PSM-5 Questionnaires | 12 weeks (± 7 days)
  Subjects' perception to medications in general measured by change from Baseline in BMQ-General-12 and PSM-5 Questionnaires at 12 weeks
Impact of mobile applications (My A:Care and Smart Coach) on the subjects' perception to medications specific to lipid-lowering therapy using BMQ-S11-Plural and MAIN Screen Questionnaires | 12 weeks (± 7 days)
  Subjects' perception to medications specific to lipid-lowering therapy measured by change from Baseline in BMQ-S11-Plural and MAIN Screen Questionnaires at 12 weeks

OTHER OUTCOMES:
Correlations between subjects' adherence to lipid-lowering therapy and mobile applications data using individual summaries retrieved from the application database. | 12 weeks (± 7 days)
  Correlations between subjects' adherence to lipid-lowering therapy and mobile applications data is measured by using individual summaries retrieved from the application database at 12 week

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pascal Berrou, MD, Phd, Study Director — Abbott
Locations (1):
- Chatlert Mueang Pongchaiyakul, Khon Kaen, Thailand

REFERENCES:
- [Derived] Pongchaiyakul C, Driessen S. Evaluating the effect of mobile applications "My A:Care" and "Smart Coach" on adherence to lipid-lowering treatment in patients with dyslipidemia: a prospective, randomized, open-label clinical study. Front Digit Health. 2025 Jul 7;7:1502990. doi: 10.3389/fdgth.2025.1502990. eCollection 2025. PMID 40692655